CLINICAL TRIAL: NCT05941507
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of TROP2-Directed Antibody-Drug Conjugate LCB84, as a Single Agent and in Combination With an Anti-PD-1 Ab, in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate TROP2 ADC LCB84 Single Agent and in Combination With an Anti-PD-1 Ab in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Collaborators: AntibodyChem Biosciences, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCB84-1001
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
Keywords: TROP2; TROP-2; Breast Cancer; Head and Neck Cancer; TNBC; Gastric Cancer; Gastroesophageal; NSCLC; Lung Cancer; Glioblastoma; Endometrial Cancer; Ovarian Cancer; Cervical Cancer; Anal Cancer; Pancreatic Cancer; Urothelial Cancer; HNSCC; Salivary gland cancer; LCB84
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Lung Neoplasms; Glioblastoma; Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Anus Neoplasms; Pancreatic Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LCB84 monotherapy (Experimental): IV infusion Q3W
  Interventions: Drug: LCB84
- LCB84 + anti-PD-1 (Experimental): IV infusion Q3W
  Interventions: Drug: LCB84; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: LCB84 — TROP2-directed human monoclonal antibody (Ab) linked to a monomethyl auristatin E (MMAE) prodrug
Drug: Anti-PD-1 monoclonal antibody — anti-PD-1 Ab
  Arms: LCB84 + anti-PD-1

SUMMARY:
This is a first-in-human, Phase 1/2 study to evaluate LCB84, a TROP2-directed antibody-drug conjugate, alone and in combination with an anti-PD-1 Ab, in dose escalation (Phase 1) followed by dose expansion (Phase 2).

The study population in dose escalation (Phase 1) consists of patients with advanced solid tumors refractory to standard of care, or for whom no standard of care exists. After the MTD and/or RP2D for single agent LCB84 is determined, dose escalation cohorts with select tumor types will be enrolled. Combination LCB84 and anti-PD-1 Ab will be evaluated in dose escalation after a minimum of 2 dose levels of single agent LCB84 have established DLT safety, to determine the MTD and/or RP2D of combination LCB84 and anti-PD-1 Ab, and to continue into dose expansion cohorts in select tumor types.

ELIGIBILITY:
Key Inclusion Criteria:

* Phase 1 Dose Escalation: histologically or cytologically confirmed advanced solid tumors refractory to standard of care treatment.
* Phase 2 Dose Expansion*: select histologically or cytologically confirmed advanced solid tumors refractory to standard of care treatment.

  *expansion cohort indications to be prioritized based on data from Phase 1 dose escalation.
* Prior treatment with TROP2-directed therapy is permitted.
* Measurable disease as defined by RECIST v1.1 or RANO-BM.
* Willingness to provide archival tumor tissue when available or to undergo pre-treatment biopsy if not available.
* Mandatory pre- and on-treatment biopsies for enrichment cohorts in Phase 1 dose escalation and Phase 2 expansion cohorts if deemed medically feasible and safe.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function as defined by:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L (1500/µL), without colony-stimulating factor support for the past 14 days
  * Platelets ≥100.0 x 109/L (100 000/µL)
  * Hemoglobin ≥9.0 g/dL
  * Aspartate aminotransferase (AST) ≤2.5 x ULN; alanine aminotransferase (ALT) ≤2.5 x ULN (AST, ALT ≤5 x ULN if liver metastases present)

Key Exclusion Criteria:

* Active or progressing central nervous system (CNS) metastases or any evidence of leptomeningeal disease.

Note: Patients with stable or treated CNS metastases may be eligible if all of the following criteria are met: 1) localized treatment for brain metastases completed at least 4 weeks prior to the first dose of study drug 2) no new or progressive neurologic symptoms and without need for immediate local therapy, steroids or anticonvulsants for symptom control (stable or decreasing steroid dose (a stable dose of ≤4 mg dexamethasone oral or equivalent) is permitted) 3) stable brain metastases for at least 1 month prior to screening (baseline) brain MRI.

* Persistent toxicities from previous systemic antineoplastic treatments >Grade 1, excluding alopecia and vitiligo.
* Systemic antineoplastic therapy (including antiestrogen therapy) within 5 half-lives or 4 weeks, whichever is shorter, prior to first dose of the study drug.
* Concomitant use of systemic steroids at dose of >10 mg of prednisone or its equivalent per day (exception for brain metastases, as described in exclusion criteria #1 above).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety of LCB84 alone and LCB84 in combination with an anti-PD-1 Ab (Phase 1 and 2) | Up to 48 months
  Incidence and severity of AEs and SAEs
Recommended Phase 2 Dose of LCB84 alone and LCB84 in combination with an anti-PD-1 Ab (Phase 1) | Up to 24 months
  Based on tolerability, preliminary anti tumor activity, and pharmacokinetics
Objective Response Rate (Phase 2) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Clinical Benefit Rate (Phase 2) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Duration of Response (Phase 2) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Time to Progression (Phase 2) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Progression Free Survival (Phase 2) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Overall Survival (Phase 2) | Up to 24 months
  Survival rates

SECONDARY OUTCOMES:
Plasma Concentrations of LCB84 (Phase 1 and 2) | Up to 48 months
  Pharmacokinetic parameters will be determined from observed concentrations of LCB84
Evaluation of the immunogenicity of LCB84 (Phase 1 and 2) | Up to 48 months
  Occurrence of ADA measured in serum at selected timepoints during the study
Objective Response Rate (Phase 1) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Duration of Response (Phase 1) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Time to Progression (Phase 1) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM
Progression Free Survival (Phase 1) | Up to 24 months
  Assessed by RECIST 1.1, iRECIST, and RANO-BM

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruiz-Soto, MD, Study Director — AntibodyChem Biosciences
Locations (8):
- United States (7):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No